CLINICAL TRIAL: NCT06846138
Title: Enhancing the Efficacy and Tolerability of Metformin by add-on Polyherbal Formulation: a Gut Microbiome Study
Acronym: Metherb
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Pauls Stradins Clinical University Hospital (Other)
Responsible Party: Principal Investigator, Valdis Pirags, Prof., Pauls Stradins Clinical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: lzp-2023/1-0422; lzp-2023/1-0422 (Other Grant/Funding Number: Latvian Council of Science)
Record Dates: First submitted 2025-02-07; First posted 2025-02-25 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus Type 2
Keywords: microbiome; metformin; diabetes; polyherbal formulation
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polyherbal formulation (Experimental): Participants in this arm will receive an add-on polyherbal formulation (PHF). Treatment Duration: 24 weeks, followed by a crossover to the placebo arm.
  Interventions: Dietary Supplement: Polyherbal Formulation (PHF); Drug: Metformin (Standard Treatment for Type 2 Diabetes)
- Placebo (Placebo Comparator): Participants in this arm will receive a placebo. Treatment Duration: 24 weeks, followed by a crossover to the PHF arm.
  Interventions: Other: Placebo; Drug: Metformin (Standard Treatment for Type 2 Diabetes)

INTERVENTIONS:
Dietary Supplement: Polyherbal Formulation (PHF) — Description: A polyherbal formulation with known beneficial effects on gut microbiota and metabolic regulation. The formulation contains selected plant extracts studied for their hypoglycemic, antioxidant, and gut microbiota-modulating properties.
  Administration: Oral, daily dosage as per study protocol. Supplier: Arya Vaidya Pharmacy (AVP), Coimbatore, India (GMP-certified).
  Arms: Polyherbal formulation
Other: Placebo — Type: Placebo Comparator Description: A placebo formulation that matches PHF in appearance, texture, and administration schedule.
  Administration: Oral, daily dosage as per study protocol.
  Arms: Placebo
Drug: Metformin (Standard Treatment for Type 2 Diabetes) — Description: Metformin is an FDA and EMA-approved antihyperglycemic medication that improves glycemic control by reducing hepatic glucose production and enhancing insulin sensitivity.
  Administration: Oral, per standard dosing guidelines. Availability: Provided to all participants per the national reimbursement scheme for T2D patients in Latvia.

SUMMARY:
Study population: Type 2 diabetes patients Design of the study: Randomized, two-arm, placebo-controlled, and prospective crossover cohort study.

Objective: To evaluate the effects of interactions between metformin and traditionally used polyherbal formulations on gut microbiota in a prospective crossover study involving type 2 diabetes mellitus patients.

Sample size: 66 patients. Duration of study: 06/2024 - 12/2026

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be eligible for enrollment:

Clinical diagnosis of Type 2 Diabetes Mellitus (T2D) HbA1c level between 6.5% and 8.5% On a stable dose of oral antidiabetic therapy for at least 6 months Age: ≥ 25 years and ≤ 80 years History of metformin intolerance, defined as previously reported gastrointestinal side effects or inability to tolerate full-dose metformin Willing and able to provide written informed consent Willing to comply with study procedures, including stool sample collection and continuous glucose monitoring (CGM)

Exclusion Criteria:

Participants will be excluded if they meet any of the following criteria:

Type 1 Diabetes Mellitus Current or recent (last 6 months) use of polyherbal formulations (PHF) Pregnancy or breastfeeding

Severe diabetic complications, such as:

Diabetic ketoacidosis Proliferative retinopathy Chronic kidney disease Stage IIIb or higher (eGFR <45 mL/min/1.73m²)

Recent cardiovascular events (within the last 6 months), including:

Stroke Myocardial infarction Unstable angina Heart failure

Severe systemic disease that could interfere with participation, such as:

Active cancer Severe autoimmune disease Current antibiotic therapy (within 2 months of study enrollment) Use of probiotics or prebiotics (within 1 month of study enrollment)

Severe gastrointestinal conditions, including:

Inflammatory bowel disease Chronic diarrhea of unknown origin Severe infection requiring antibacterial therapy Participation in another interventional study within the last 3 months

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Glycemic Control (HbA1c Levels) | Baseline, Week 24, Week 48
  Measurement of HbA1c (%) to evaluate the impact of PHF on glycemic control compared to placebo.

SECONDARY OUTCOMES:
Relative Abundance of Key Bacterial Taxa in Gut Microbiota | Baseline, Week 2, Week 24, Week 25, Week 48
  Description: Measurement of the relative abundance of specific bacterial taxa (Akkermansia muciniphila, Escherichia spp., Intestinibacter) in fecal samples using metagenomic sequencing.
Gastrointestinal Tolerability of Metformin | Baseline, Week 2, Week 24, Week 25, Week 48
  Assessment of gastrointestinal side effects, including nausea, bloating, diarrhea, and abdominal discomfort, using a standardized gut microbiota-related symptom questionnaire.
  Scale Name: Gastrointestinal Symptom Rating Scale (GSRS) Score Range: Minimum = 0, Maximum = 4 Interpretation: Lower scores indicate better gastrointestinal tolerability.
Fasting and Postprandial Blood Glucose Levels | Baseline, Week 24, Week 48
  Measurement of fasting and postprandial glucose levels using standard biochemical assays.
  Unit of Measure: mmol/L
Time in Range (TIR) Measured by Continuous Glucose Monitoring (CGM) | Week 1
  Time in Range (TIR) Measured by Continuous Glucose Monitoring (CGM) Description: Measurement of the percentage of time that blood glucose levels remain within the target range (70-180 mg/dL) using data from Continuous Glucose Monitoring (CGM).
Metabolomic Analysis of Stool Samples (Short-chain fatty acids (SCFAs)) | Baseline, Week 24, Week 48
  The levels of acetic acid, propionic acid, isobutyric acid, butyric acid, isovaleric acid, valeric acid, and caproic acid will be quantified using gas chromatography-mass spectrometry (GC-MS). These concentrations will be reported in micromoles per gram of fecal matter (μmol/g).
Patient-Reported Outcomes on Quality of Life | Baseline, Week 24, Week 48
  Description: Evaluation using a validated diabetes-related quality of life questionnaire. Diabetes Quality of Life (DQOL) Questionnaire.
  Scoring: Items are scored on a 5-point Likert scale, with higher scores typically indicating more negative impacts or dissatisfaction.
Metabolomic Analysis of Stool Samples (Amino acids) | Baseline, Week 24, Week 48
  The following amino acids will be analyzed using ultra-high-performance liquid chromatography-mass spectrometry (UHPLC-MS): acetylcarnitine, arginine, butyrylcarnitine, carnitine, citrulline, creatinine, glutamic acid, glutamine, histidine, isoleucine, leucine, lysine, methionine, ornithine, phenylalanine, proline, serotonin, taurine, tryptophan, tyrosine, and valine. Results will be expressed in nanomoles per gram of fecal matter (nmol/g).
Metabolomic Analysis of Stool Samples (Bile acids) | Baseline, Week 24, Week 48
  The bile acids to be measured include cholic acid, chenodeoxycholic acid, deoxycholic acid, and lithocholic acid, along with their conjugated forms: glycocholic acid, glycochenodeoxycholic acid, glycodeoxycholic acid, glycolithocholic acid, taurocholic acid, taurochenodeoxycholic acid, taurodeoxycholic acid, taurolithocholic acid, and ursodeoxycholic acid. These will be quantified using liquid chromatography-mass spectrometry (LC-MS), with concentrations reported in micromoles per gram of fecal matter (μmol/g).

CONTACTS AND LOCATIONS:
Locations (1):
- Pauls Stradins Clinical University Hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF